CLINICAL TRIAL: NCT07387861
Title: Immunohistochemical Evaluation of p-AKT and p-S6 as Surrogate Markers of PI3K/AKT/mTOR Pathway Activation in ER-Positive, HER2-Negative Breast Carcinoma
Brief Title: PI3K Pathway Activation Markers in ER-Positive, HER2-Negative Breast Cancer: A Clinicopathologic Study
Acronym: p-AKT p-S6
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Roaa Ahmed Mohamed Elnaffar, Demonstrator, Assiut University
Other Study IDs: Pending
Record Dates: First submitted 2026-01-25; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer - ER+, HER2-, PIK3CA Gene Mutation
Keywords: Breast Cancer; PI3K/AKT/mTOR pathway; Phospho-AKT; Phospho-S6; Endocrine therapy; Tumor budding; TILs
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endocrine-Resistant Breast Cancer: Patients with ER-positive, HER2-negative invasive breast carcinoma who developed primary or secondary resistance to adjuvant endocrine therapy.
  Interventions: Other: Not applicable- observational study
- Endocrine-Sensitive Breast Cancer: Patients with ER-positive, HER2-negative invasive breast carcinoma who remained relapse-free during adjuvant endocrine therapy and for ≥12 months after completion, with sufficient follow-up.
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — Not Applicable. This is an observational study; no interventions are assigned.

SUMMARY:
The goal of this observational study is to examine whether markers of PI3K pathway activation are associated with endocrine therapy response and clinicopathologic features in estrogen receptor-positive, HER2-negative breast cancer. The main questions it aims to answer are:

Are immunohistochemical levels of phosphorylated AKT (p-AKT) and phosphorylated S6 (p-S6) different between endocrine-sensitive and endocrine-resistant breast cancer cases? Do different levels of p-AKT and p-S6 show distinct clinicopathologic and histologic characteristics, including features of the tumor microenvironment?

Archived tumor tissue from patients who received adjuvant endocrine therapy as part of routine clinical care will be analyzed. Biomarker expression will be correlated with clinicopathologic parameters, including tumor-infiltrating lymphocyte density, tumor budding, and other histologic features, to explore associations with tumor behavior and outcomes.

DETAILED DESCRIPTION:
Endocrine therapy is the cornerstone of treatment for estrogen receptor-positive breast cancer; however, a substantial proportion of patients develop resistance during the disease course. Activation of the PI3K/AKT/mTOR signaling pathway has been implicated as a key mechanism underlying resistance to endocrine therapy and disease progression. While genomic alterations in PI3K pathway-related genes are commonly assessed, they do not consistently reflect pathway activation or predict therapeutic response, highlighting the need for practical surrogate biomarkers.

The aim of this study is to evaluate immunohistochemical markers of PI3K pathway activation in estrogen receptor-positive, HER2-negative invasive breast carcinoma and to explore their associations with endocrine therapy response and clinicopathologic characteristics. Specifically, the study examines whether levels of phosphorylated AKT (p-AKT) and phosphorylated S6 (p-S6) differ between endocrine-sensitive and endocrine-resistant cases and whether these markers correlate with histologic features related to tumor biology and the tumor microenvironment.

This is a retrospective observational study including patients with estrogen receptor-positive, HER2-negative invasive breast carcinoma who received adjuvant endocrine therapy as part of routine clinical care. Archived formalin-fixed, paraffin-embedded (FFPE) tissue blocks from excisional surgical specimens will be retrieved, and clinicopathologic and follow-up data will be collected from medical records.

Cases will be classified into endocrine-sensitive and endocrine-resistant groups based on international consensus definitions using the timing of disease recurrence relative to endocrine therapy. Immunohistochemical staining for p-AKT and p-S6 will be performed on FFPE tissue sections and evaluated using a semi-quantitative scoring system. Histopathologic assessment will include standard reporting parameters as well as additional features such as tumor-infiltrating lymphocyte density, tumor budding, lymphovascular invasion, perineural invasion, and tumoral necrosis. Associations between biomarker expression, clinicopathologic features, and follow-up outcomes will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with invasive breast carcinoma.
* ER-positive and HER2-negative tumor status.
* Received adjuvant endocrine therapy as part of routine clinical care.
* Archived formalin-fixed paraffin-embedded (FFPE) tumor tissue available from excisional specimens (mastectomy).
* Available medical records documenting treatment history and follow-up outcomes.

Exclusion Criteria:

* Cases with missing or unavailable FFPE tissue blocks.
* Cases with insufficient tissue quality for immunohistochemistry (e.g., severely degraded or exhausted FFPE block).
* Cases with unknown or incomplete follow-up or treatment data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with estrogen receptor-positive (ER+), HER2-negative invasive breast cancer who received adjuvant endocrine therapy and have available formalin-fixed, paraffin-embedded (FFPE) tumor tissue archived in the Surgical Pathology Laboratory of Assiut University Hospital, as well as corresponding clinical follow-up data in the medical records of the Oncology Department at Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Immunohistochemical expression of PI3K pathway activation markers: p-AKT and p-S6. | At the time of immunohistochemical staining of archived tissue (single time point).
  Semi-quantitative assessment of phosphorylated AKT (Ser473) and phosphorylated S6 ribosomal protein in FFPE breast carcinoma tissue sections, scored using H-score, to compare expression levels between endocrine-sensitive and endocrine-resistant ER-positive, HER2-negative cases.

SECONDARY OUTCOMES:
Correlation of p-AKT and p-S6 expression with endocrine therapy response. | through study completion, an average of 2 years
  Description: Association of biomarker expression with endocrine therapy response (sensitive vs resistant) and time to recurrence or progression.
Correlation of p-AKT and p-S6 expression with histologic features | through study completion, an average of 2 years
  Association of biomarker expression with tumor grade, histologic type, luminal subtype, tumor budding, tumor-infiltrating lymphocyte (TIL) density, lymphovascular invasion, perineural invasion, and tumor necrosis.
Correlation of p-AKT and p-S6 expression with clinicopathologic features | through study completion, an average of 2 years
  Description: Association of biomarker expression with patient age, menopausal status, tumor size, nodal status, and stage at presentation.

CONTACTS AND LOCATIONS:
Overall Officials: Roaa A Elnaffar, MBBS, Principal Investigator — Assiut University, Faculty of Medicine

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant-level data will not be publicly shared because the study uses archived clinical and pathology records containing sensitive patient information. Although the data will be de-identified, sharing it broadly could risk patient privacy and confidentiality. Data may be shared on a case-by-case basis with qualified researchers after institutional review and approval.

REFERENCES:
- [Background] Lv W, Du C, Zhang Y, Wu F, Jin Y, Chen X, Liu X, Feng C, Ma X, Zhang S. Clinicopathological characteristics and prognostic analysis of PIK3CA mutation in breast cancer patients in Northwest China. Pathol Res Pract. 2022 Oct;238:154063. doi: 10.1016/j.prp.2022.154063. Epub 2022 Aug 10. PMID 35994807
- [Background] Adamo B, Deal AM, Burrows E, Geradts J, Hamilton E, Blackwell KL, Livasy C, Fritchie K, Prat A, Harrell JC, Ewend MG, Carey LA, Miller CR, Anders CK. Phosphatidylinositol 3-kinase pathway activation in breast cancer brain metastases. Breast Cancer Res. 2011;13(6):R125. doi: 10.1186/bcr3071. Epub 2011 Dec 1. PMID 22132754
- [Background] Maruyama N, Miyoshi Y, Taguchi T, Tamaki Y, Monden M, Noguchi S. Clinicopathologic analysis of breast cancers with PIK3CA mutations in Japanese women. Clin Cancer Res. 2007 Jan 15;13(2 Pt 1):408-14. doi: 10.1158/1078-0432.CCR-06-0267. Epub 2007 Jan 3. PMID 17202311
- [Background] Sakr RA, Weigelt B, Chandarlapaty S, Andrade VP, Guerini-Rocco E, Giri D, Ng CK, Cowell CF, Rosen N, Reis-Filho JS, King TA. PI3K pathway activation in high-grade ductal carcinoma in situ--implications for progression to invasive breast carcinoma. Clin Cancer Res. 2014 May 1;20(9):2326-37. doi: 10.1158/1078-0432.CCR-13-2267. Epub 2014 Mar 14. PMID 24634376
- [Background] Rasti AR, Guimaraes-Young A, Datko F, Borges VF, Aisner DL, Shagisultanova E. PIK3CA Mutations Drive Therapeutic Resistance in Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer. JCO Precis Oncol. 2022 Mar;6:e2100370. doi: 10.1200/PO.21.00370. PMID 35357905
- [Background] Pierobon M, Ramos C, Wong S, Hodge KA, Aldrich J, Byron S, Anthony SP, Robert NJ, Northfelt DW, Jahanzeb M, Vocila L, Wulfkuhle J, Gambara G, Gallagher RI, Dunetz B, Hoke N, Dong T, Craig DW, Cristofanilli M, Leyland-Jones B, Liotta LA, O'Shaughnessy JA, Carpten JD, Petricoin EF. Enrichment of PI3K-AKT-mTOR Pathway Activation in Hepatic Metastases from Breast Cancer. Clin Cancer Res. 2017 Aug 15;23(16):4919-4928. doi: 10.1158/1078-0432.CCR-16-2656. Epub 2017 Apr 26. PMID 28446508
- [Background] Creighton CJ, Fu X, Hennessy BT, Casa AJ, Zhang Y, Gonzalez-Angulo AM, Lluch A, Gray JW, Brown PH, Hilsenbeck SG, Osborne CK, Mills GB, Lee AV, Schiff R. Proteomic and transcriptomic profiling reveals a link between the PI3K pathway and lower estrogen-receptor (ER) levels and activity in ER+ breast cancer. Breast Cancer Res. 2010;12(3):R40. doi: 10.1186/bcr2594. Epub 2010 Jun 22. PMID 20569503
- [Background] Cascardo F, Vivanco M, Perrone MC, Werbach A, Enrico D, Mando P, Amat M, Martinez-Vazquez P, Burruchaga J, Mac Donnell M, Lanari C, Zwenger A, Waisberg F, Novaro V. Higher risk of recurrence in early-stage breast cancer patients with increased levels of ribosomal protein S6. Sci Rep. 2024 Oct 24;14(1):25136. doi: 10.1038/s41598-024-75154-1. PMID 39448637
- [Background] Miller TW, Rexer BN, Garrett JT, Arteaga CL. Mutations in the phosphatidylinositol 3-kinase pathway: role in tumor progression and therapeutic implications in breast cancer. Breast Cancer Res. 2011;13(6):224. doi: 10.1186/bcr3039. Epub 2011 Nov 1. PMID 22114931
- [Background] Skolariki A, D'Costa J, Little M, Lord S. Role of PI3K/Akt/mTOR pathway in mediating endocrine resistance: concept to clinic. Explor Target Antitumor Ther. 2022;3(2):172-199. doi: 10.37349/etat.2022.00078. Epub 2022 Apr 24. PMID 36046843
- [Background] Toska E, Osmanbeyoglu HU, Castel P, Chan C, Hendrickson RC, Elkabets M, Dickler MN, Scaltriti M, Leslie CS, Armstrong SA, Baselga J. PI3K pathway regulates ER-dependent transcription in breast cancer through the epigenetic regulator KMT2D. Science. 2017 Mar 24;355(6331):1324-1330. doi: 10.1126/science.aah6893. Erratum In: Science. 2019 Jan 25;363(6425):eaaw7574. doi: 10.1126/science.aaw7574. PMID 28336670
- [Background] Vasan N, Toska E, Scaltriti M. Overview of the relevance of PI3K pathway in HR-positive breast cancer. Ann Oncol. 2019 Dec 1;30(Suppl_10):x3-x11. doi: 10.1093/annonc/mdz281. PMID 31859348
- [Background] Lei JT, Anurag M, Haricharan S, Gou X, Ellis MJ. Endocrine therapy resistance: new insights. Breast. 2019 Nov;48 Suppl 1(Suppl 1):S26-S30. doi: 10.1016/S0960-9776(19)31118-X. PMID 31839155
- [Background] Hanker AB, Sudhan DR, Arteaga CL. Overcoming Endocrine Resistance in Breast Cancer. Cancer Cell. 2020 Apr 13;37(4):496-513. doi: 10.1016/j.ccell.2020.03.009. PMID 32289273